CLINICAL TRIAL: NCT04749589
Title: Fatigue, Quality of Life, Cognitive Function and Physical Ability in Patients Suspected of Colorectal Malignancy
Status: Completed | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 21 6250
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Colorectal Cancer; Fatigue; Quality of Life; Cognitive Impairment
MeSH Terms: conditions — Anemia, Iron-Deficiency; Colorectal Neoplasms; Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iron deficient: ferritin<30 or Transferine saturation<.2
  Interventions: Diagnostic Test: iron deficiency
- iron replete: opposite of the other group
  Interventions: Diagnostic Test: iron deficiency

INTERVENTIONS:
Diagnostic Test: iron deficiency — Its not an intervention. Its an observational study. The groups are defined based on their iron status

SUMMARY:
The aim is to investigate if iron deficiency at the time of colorectal cancer diagnosis has an influence on fatigue, quality of life, cognition and physical ability.

DETAILED DESCRIPTION:
Around 60% of newly diagnosed colorectal cancer patients suffer from iron deficiency at the time of diagnosis. The study hypothesis is that, besides leading to anemia, iron deficiency might be associated with impaired patient report outcomes in the domains of fatigue, quality of life, cognitive impairment and lower physical ability. No previous studies on colorectal cancer patients and iron deficiency are available.

The participants (patients suspected of colorectal cancer after endoscopy) will be tested on these parameters. The participants and the investigators are blinded to the patients iron status. The study takes place before any preoperative iron treatment. Multivariate analysis will be used taking into account, gender, age, hemoglobin, tumor stage.

ELIGIBILITY:
Inclusion Criteria:

* patients in whom endoscopy has raised suspicion of colorectal malignancy

Exclusion Criteria:

* non fluent in Danish language
* cerebral impairment (ex severe dementia) so that informed consent can not be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see inclusion criteria
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Fatigue | up to one months after inclusion
  Fatigue sub-scale of Focussed assessment of cancer treatment - anemia

SECONDARY OUTCOMES:
Quality of life | up to one months after inclusion
  European Organisation for Research and Treatment of Cancer C30
Cognitive ability | up to one months after inclusion
  Montreal cognitive assessment
endurance | up to one months after inclusion
  6 minutes walk test
peripheral muscular strengths | up to one months after inclusion
  hand-held dynamometer
mobility and balance | up to one months after inclusion
  timed-up-and-go-test

OTHER OUTCOMES:
post-operative run | 30-days postoperatively
  the ability of the above mentioned test to predict the postoperative run (complications/length of stay)

CONTACTS AND LOCATIONS:
Overall Officials: Torben Knudsen, ass. prof, Study Director — Institute of regional health research, regional of southern denmark
Locations (3):
- Denmark (3):
  - Sygehus Sønderjylland, Aabenraa, Region Syddanmark
  - Hospital of South West Jutland, Esbjerg, Region Syddanmark
  - Hospital of South West Jutland, Grindsted, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No